CLINICAL TRIAL: NCT06856642
Title: Comparison of Abdominal Draw-in Maneuver With Real-time Ultrasound Imaging Biofeedback vs Conservative Physical Therapy in Patients With Chronic Low Back Pain: A Prospective, Randomized Clinical Trial
Brief Title: Comparison of Abdominal Draw-in Maneuver With Real-time Ultrasound Imaging Biofeedback vs Conservative Physical Therapy in Patients With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-09
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: chronic non-specific low back pain; low back pain; ultrasound imaging; real-time ultrasound biofeedback; biofeedback; abdominal draw-in manuever
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-Time Ultrasound Biofeedback with Abdominal Draw-In Manuever (Active Comparator)
  Interventions: Other: Conservative Physical Therapy; Other: Real-Time Ultrasound Biofeedback with Abdominal Draw-In Manuever
- Conservative treatment group without biofeedback (Active Comparator)
  Interventions: Other: Conservative Physical Therapy; Other: Abdominal Draw-in Manuever

INTERVENTIONS:
Other: Conservative Physical Therapy — Transcutaneous Electrical Nerve Stimulation (TENS):It is an electrotherapy modality commonly used in pain management. Conventional TENS will be applied to our patients. The frequency of Conventional TENS will be 50 Hz, the pulse duration will be 80 µs, the amplitude will be of mild to moderate intensity as perceived by the patient, and the duration will be 20 minutes.
  Hot Pack:It is a superficial heat therapy method commonly used to reduce muscle spasms, increase circulation, and alleviate pain.The packs, which are kept in hydrocollator tanks, will be applied at a temperature that will not harm the patient.The application time is 20 minutes.
  Therapeutic Ultrasound:This method, which uses sound waves to support tissue healing, creates heating and healing effects in deep tissues and is commonly used to reduce pain and relieve muscle spasmsThe frequency of the applied ultrasound will be 1 MHz, with an intensity of 1.5 W/cm², and it will be applied for 8 minutes in continuous mode
Other: Abdominal Draw-in Manuever — Starting Position: The patient lies in a supine position with knees bent and feet flat on the ground. The neck and spine are kept in a neutral position. Breath Control: The patient focuses on abdominal expansion while inhaling and flattening the abdomen while exhaling. Transversus Abdominis Activation: The patient attempts to draw the abdominal muscles inward (pulling the navel toward the spine). During this movement, care should be taken to avoid pressing the lower back against the ground or contracting the hip muscles. The goal is to activate only the deep abdominal muscles. Checking for Proper Muscle Activation: The patient can place their fingertips on the lower abdominal region (just above the pelvic bone) to feel whether the transversus abdominis muscle is activating correctly. Maintaining the Position: The patient holds this activation for 5-10 seconds while continuing to breathe naturally, then relaxes. Muscles should be fully relaxed between repetitions.
  Arms: Conservative treatment group without biofeedback
Other: Real-Time Ultrasound Biofeedback with Abdominal Draw-In Manuever — The patient, who has been instructed on the abdominal drawing-in exercise, assumes a supine position with knees bent. The ultrasound screen is positioned so that both the practitioner and the patient can see it. The researcher places the linear ultrasound probe on the patient's transversus abdominis muscle to obtain an image, which is then shown to the patient for awareness. The patient is instructed to keep their eyes on the screen and follow their muscle activity throughout the exercise. During the exercise, the patient's muscle is displayed on the screen, and they are asked to hold the contraction at its maximum level for 10 seconds. After the contraction phase, the patient is instructed to relax and rest for 2 minutes. The treatment is completed with a total of 10 repetitions.
  Arms: Real-Time Ultrasound Biofeedback with Abdominal Draw-In Manuever

SUMMARY:
The aim of this study is to compare the effectiveness of abdominal drawing-in maneuver with real-time ultrasound biofeedback to conservative treatment in patients with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Low back pain is a common clinical condition among musculoskeletal disorders. It can be classified into two main categories: acute and chronic. Acute low back pain is usually limited to a duration of 6 weeks or less, whereas chronic low back pain refers to pain lasting 12 weeks or longer. Chronic low back pain is characterized by persistent and untreated pain, which can significantly affect individuals' physical and psychological health. A multidisciplinary approach is required for its treatment. Physical therapy, pharmacological approaches, psychotherapy, and exercise are the main treatment methods.

Exercise plays an active role in both the prevention and treatment of the disease. Among many exercise methods, the abdominal drawing-in maneuver has been proven effective in the literature. Biofeedback is a technique that helps individuals consciously control their physiological processes. Real-time ultrasound biofeedback stands out as a technique that directly visualizes musculoskeletal system functions. This method uses high-frequency sound waves to assess the dynamic movements of internal organs and muscle structures. Through this technology, individuals can visualize their movements in real time and consciously adjust their muscle activity or posture. It offers significant advantages, particularly in clinical and sports applications such as pelvic floor rehabilitation, postural balance training, and motor control skill development.

The aim of our study is to compare the effectiveness of exercises performed with real-time ultrasound biofeedback with those in patients receiving conservative treatment. Patients will be randomly assigned to two groups: Group 1: Patients receiving conservative treatment and performing the abdominal drawing-in maneuver with real-time ultrasound imaging biofeedback. Group 2 (Control Group): Patients receiving conservative treatment and performing the abdominal drawing-in maneuver with only verbal instruction. A total of 40 patients are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* The duration of low back pain is at least 3 months.
* Low back pain with or without radiation to the lower extremities.
* Age between 18-65 years.
* Chronic nonspecific low back pain patients.

Exclusion Criteria:

* Neuropathic pain complaints.
* Pregnancy status.
* History of infection, cancer, or trauma.
* Neurological abnormalities.
* History of lumbar spine surgery.
* History of conservative physical therapy and/or injections in the lumbar region within the last 6 months.
* Neurological diseases such as Parkinson's or Multiple Sclerosis.
* Systemic diseases that prevent exercise.
* Patients with a Mini-Mental Test score below 24.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | before treatment
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Visual Analogue Scale | In the 3rd week of treatment
  Pain was evaluated using a 10 cm long Visual Analogue Scale (VAS) during rest and activity (0 = no pain, 10 = very severe pain).
Muscle Thickness | before treatment
  The linear probe is placed transversely at the point where the iliac crest intersects with the middle point of the T12 rib, crossing the mid-axillary line. The position of the linear probe is adjusted until all abdominal muscles are visible. To standardize the images, the center point of the probe in the image is shifted 2 cm laterally to align with the insertion of the superficial fascia of the transversus abdominis muscle. The thickness of the transversus abdominis muscle is determined by the distance between the superficial and deep fascia at the thickest point in the image. The thickness between the two fasciae is measured using the digital caliper of the device.
Muscle Thickness | In the 3rd week of treatment
  The linear probe is placed transversely at the point where the iliac crest intersects with the middle point of the T12 rib, crossing the mid-axillary line. The position of the linear probe is adjusted until all abdominal muscles are visible. To standardize the images, the center point of the probe in the image is shifted 2 cm laterally to align with the insertion of the superficial fascia of the transversus abdominis muscle. The thickness of the transversus abdominis muscle is determined by the distance between the superficial and deep fascia at the thickest point in the image. The thickness between the two fasciae is measured using the digital caliper of the device.

SECONDARY OUTCOMES:
Berg Balance Scale | before treatment
  The Berg Balance Scale is an assessment tool developed to measure balance performance in geriatric patients. It is frequently used in clinical studies to evaluate postural control and predict fall risk. The scale consists of 14 instructions, and the patient's performance for each instruction is observed and scored from 0 to 4. A score of 0 is given when the patient is unable to perform the activity at all, while a score of 4 is given when the patient completes the activity independently.
Berg Balance Scale | In the 3rd week of treatment
  The Berg Balance Scale is an assessment tool developed to measure balance performance in geriatric patients. It is frequently used in clinical studies to evaluate postural control and predict fall risk. The scale consists of 14 instructions, and the patient's performance for each instruction is observed and scored from 0 to 4. A score of 0 is given when the patient is unable to perform the activity at all, while a score of 4 is given when the patient completes the activity independently.
Oswestry Disability Index | before treatment
  The Oswestry Disability Index is a specific questionnaire method used to assess functional status in patients with low back pain. It consists of 10 items, each evaluating the impact of low back pain on daily living activities. Each item is rated from 0 to 5, and the total score is converted into a percentage for evaluation. A total score of 0-20%: Minimal disability, 21-40%: Moderate disability, 41-60%: Severe disability, 61-80%: Crippled condition, and 81-100%: Complete disability.
Oswestry Disability Index | In the 3rd week of treatment
  The Oswestry Disability Index is a specific questionnaire method used to assess functional status in patients with low back pain. It consists of 10 items, each evaluating the impact of low back pain on daily living activities. Each item is rated from 0 to 5, and the total score is converted into a percentage for evaluation. A total score of 0-20%: Minimal disability, 21-40%: Moderate disability, 41-60%: Severe disability, 61-80%: Crippled condition, and 81-100%: Complete disability.
Lomber Range of Motion | before treatment
  The range of motion of lomber region will be measured passively with a goniometer in the flexion, abduction, internal rotation and external rotation directions.
Lomber Range of Motion | In the 3rd week of treatment
  The range of motion of lomber region will be measured passively with a goniometer in the flexion, abduction, internal rotation and external rotation directions.
EQ-5D-3L General Quality of Life Scale | before treatment
  The EQ-5D-3L is a standardized, simple, and short questionnaire method used to measure individuals' overall health status. It contains five questions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. For each question, a 3-level assessment is made (1: No problems, 2: Moderate problems, 3: Severe problems).
EQ-5D-3L General Quality of Life Scale | In the 3rd week of treatment
  The EQ-5D-3L is a standardized, simple, and short questionnaire method used to measure individuals' overall health status. It contains five questions: mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. For each question, a 3-level assessment is made (1: No problems, 2: Moderate problems, 3: Severe problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)